CLINICAL TRIAL: NCT06758115
Title: Study on the Central Motor Regulation Mechanism in Adolescent Idiopathic Scoliosis (AIS) Patients Based on HD-sEMG, EEG, and Neuromuscular Coupling Analysis
Brief Title: Central Motor Mechanisms in AIS Via HD-sEMG, EEG and Neuromuscular Coupling Analysis
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KL-504-02
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Massage; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIS
  Interventions: Procedure: Tuina (Massage) Therapy
- Healthy Control Group
  Interventions: Procedure: Tuina (Massage) Therapy

INTERVENTIONS:
Procedure: Tuina (Massage) Therapy — Operation Method:
  Correct abnormal joint alignment - Manipulatively realign the vertebral segments and pelvis affected by scoliosis.
  Correct abnormal muscle function - After realigning the vertebral bodies to their normal position, stretch the corresponding tight and shortened muscles while strengthening the muscles that need to be lengthened.
  Restore joint stability - After adjusting the vertebrae and muscles, instruct the patient to hold the corrected posture for at least 10 seconds, then relax for 10 seconds. Repeat this cycle 3-5 times.
  Restore sensorimotor control - Provide appropriate movement disturbances to patients maintaining the corrected posture to enhance proprioception and motor memory in the corresponding muscles.
  The total duration of the manipulation is 20-25 minutes. Treatment is performed twice a week for a total of 12 weeks.

SUMMARY:
1. Verifying the Motor Control Effects of Spinal Manipulation on AIS Using outpatient and inpatient AIS patients from our department as the study subjects, standardized spinal manipulation treatment is applied. The efficacy is evaluated through a combination of clinical outcome measures, HD-EMG for paraspinal muscle function assessment, and Pro-Kin balance system for trunk stability analysis. This establishes an AIS efficacy platform to further clarify the effectiveness of spinal manipulation in motor control regulation of AIS.
2. Investigating the Central Motor Network's Response to Spinal Manipulation in AIS Utilizing high-density sEMG-EEG technology, synchronized brain and muscle electrical signals are collected before and after treatment. By employing a neuromuscular synchronization and coupling analysis approach that integrates linear and nonlinear methods, the characteristic indices of information interaction between the central system and muscles are identified. This further explores the motor control and response characteristics of the muscle-cortex network to spinal manipulation in AIS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥10 years;
2. Risser sign grade 0-3;
3. Cobb angle between 10° and 40°;
4. No prior treatment;
5. Female patients within 1 year after menarche or before menstruation;
6. The patient's guardian signs the informed consent form for treatment.

Exclusion Criteria:

1. Those who do not meet the diagnostic criteria for AIS or inclusion criteria;
2. Patients with severe primary diseases such as cardiovascular, cerebrovascular, liver, kidney, and hematopoietic system disorders, or those with mental illnesses;
3. Patients with thrombocytopenia, coagulation disorders, or a tendency to bleed;
4. Patients who are afraid of the treatment and cannot tolerate it;
5. Those who have already received other treatments that may affect the study's outcome measures.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent Idiopathic Scoliosis Patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HD-EMG | Before treatment, and at 4 weeks and 12 weeks after treatment.
  Muscle performance was assessed using the SAGA high-density electromyography (EMG) system to evaluate the function and activity of the paraspinal muscles.

SECONDARY OUTCOMES:
Pro-Kin Balance System | Before treatment, and at 4 weeks and 12 weeks after treatment.
  The Pro-Kin Balance System was used to assess trunk stability and evaluate motor control ability.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No